CLINICAL TRIAL: NCT01862666
Title: A Comparison of Volumetric Laser Endomicroscopy (VLE) and Endoscopic Mucosal Resection (EMR) in Patients With Barrett's Dysplasia or Intramucosal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: NinePoint Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 12_01
Record Dates: First submitted 2013-05-16; First posted 2013-05-24 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2014-03

CONDITIONS: Barrett'S-associated Dysplasia; Intramucosal Adenocarcinoma
Keywords: Barrett's Esophagus; Dysplasia; Intramucosal Adenocarcinoma; EMR; Endoscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endoscopic Mucosal Resection (EMR). With this technique, the mucosa is resected by injecting a liquid in the submucosal space, after which the thus created pseudopolyp can be resected using a snare and electrocoagulation. The histological processing of the ex-vivo EMR specimen will be carried out according to hospital standards
Oversight: Data Monitoring Committee: No

SUMMARY:
Barrett's esophagus (BE) is a pre-neoplastic condition formed by the metaplasia of the normal squamous mucosa of the distal esophagus into a specialized intestinal mucosa. Its development is mostly associated with chronic injury from gastroesophageal reflux. BE is widely considered the leading risk factor for the development of esophageal adenocarcinoma (EAC).

Volumetric laser endomicroscopy (VLE) can be thought of as an analogous technique to ultrasound, however, instead of producing an image from the scattering of sound waves, it utilizes optical scattering based on differences in tissue composition to form a two-dimensional image. The benefit of VLE over ultrasound is that it is capable of generating cross-sectional images of tissues with an axial-resolution of up to 10 micrometers, which is comparable to low-power microscopy.

The proposed trial will evaluate the ability of physicians to use VLE to visualize high grade intraepithelial neoplasia (HGIN) or intramucosal adenocarcinoma (IMC) in both the ex-vivo and in-vivo setting and correlate those images to standard histology of endoscopic mucosal resection specimens as the gold standard.

DETAILED DESCRIPTION:
The diagnosis of dysplasia and early adenocarcinoma in BE remains challenging. At present, endoscopy with biopsy of suspected BE lesions is the only available method. However, the endoscopic recognition of early dysplasia in BE relies on the subjective visual recognition by an endoscopist. The subtle mucosal variations and early dysplastic changes in the esophagus may easily be missed. The development of a wide-field, high resolution endoscopic microscopy could enhance the early detection and treatment of dysplasia in BE.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 years.
* Patients with either suspected or confirmed Barrett's-associated dysplasia or intramucosal adenocarcinoma presenting for endoscopy likely requiring EMR.

  - Only en-bloc resections will be investigated, requiring lesions with a maximum diameter of 15 mm with a Paris classification of 0-IIa, b, c, or a combination.
* Ability to provide written, informed consent.
* Women of childbearing potential must be willing to take a pregnancy test.

Exclusion Criteria:

* Patients on anticoagulation.
* Patients with esophageal varices that preclude either mucosal resection or biopsies.
* Presence of an esophageal mass that precludes full distention of the balloon from the NvisionVLE Catheter.
* Patients with esophageal strictures that would prevent adequate expansion of the balloon from the NvisionVLE Catheter.
* Patients with known inflammatory disease, esophageal tears or ulcers, which would prohibit full distention of the balloon from the NvisionVLE Catheter.
* Patients with known eosinophilic esophagitis.
* Patients that are pregnant.
* Patients with a history of hemostasis disorders*.
* Patients with esophagitis above grade A.

  * Hemostasis disorders will include, but will not be limited to: patients with hemophilia or other congenitally acquired clotting factor deficiencies, patients with cirrhosis with coagulopathy, patients known to have thrombocytopenia (<100,000 plt/ul) and individuals with von Willibrand's disease or other known platelet malfunction disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either suspected or confirmed Barrett's-associated dysplasia or intramucosal adenocarcinoma presenting for endoscopy likely requiring EMR.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The correlation of features seen on VLE images to those seen on histopathology from mucosal resection specimens. | VLE images will be obtained during the day of the EGD (baseline). There is no follow-up period for this protocol. Correlation of features from VLE to histo will occur at the completion of enrollment.
  All VLE images will be evaluated by two independent reviewers (not the trial endoscopist performing the scan), who are blinded to the histological finding of the corresponding EMR specimen. A predefined classification scheme will be used for VLE assessment.

SECONDARY OUTCOMES:
The creation of an image atlas, to determine the intra- and inter-observer agreement on VLE images in correlation with histopathology, resulting in refinement of the existing VLE image interpretation criteria and the validation of the VLE classification. | VLE images will be obtained during the day of the EGD (baseline). There is no follow-up period for this protocol. The creation of the image atlas will occur at the completion of enrollment.
  All VLE images will be evaluated by two independent reviewers (not the trial endoscopist performing the scan), who are blinded to the histological finding of the corresponding EMR specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Bergman, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, AZ, Netherlands

REFERENCES:
- [Derived] Swager AF, Tearney GJ, Leggett CL, van Oijen MGH, Meijer SL, Weusten BL, Curvers WL, Bergman JJGHM. Identification of volumetric laser endomicroscopy features predictive for early neoplasia in Barrett's esophagus using high-quality histological correlation. Gastrointest Endosc. 2017 May;85(5):918-926.e7. doi: 10.1016/j.gie.2016.09.012. Epub 2016 Sep 19. PMID 27658906